CLINICAL TRIAL: NCT05952310
Title: Multicenter, Open-label, Phase I/II Clinical Trial of Infusion of Activated NK Cells for the Treatment of Children, Adolescents and Young Adults With Sarcomas
Brief Title: Clinical Trial of Infusion of Activated NK Cells for the Treatment of Sarcomas
Acronym: SANKOMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Pérez Martínez (Other)
Responsible Party: Sponsor-Investigator, Antonio Pérez Martínez, Chief of Pediatric Hemato-Oncology and Hematopoietic Transplantation Service, Instituto de Investigación Hospital Universitario La Paz
Organization: Instituto de Investigación Hospital Universitario La Paz (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SANKOMA_2016
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Malignant Sarcoma
MeSH Terms: interventions — Cell Count

STUDY DESIGN:
Intervention Model Description: This is an exploratory, open-label, non-randomized, multicenter therapeutic study. It is considered phase I/II since it will seek safety and efficacy of the infusion of allogeneic haploidentical Natural Killer (NK) cells in combination with chemotherapy and/or radiotherapy in the treatment of pediatric, adolescent and young adult patients with refractory sarcoma.
Masking Description: There is no masking in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic Natural Killer cells (Experimental): Low doses (1x106/UI/m2) of subcutaneous interleukin-2 (IL-2) will be administered every 48h for a maximum of 6 doses, in conjunction with the NK cell infusion, to favor the expansion and antitumor effect of the NK cells.
  Interventions: Other: Natural Killer (NK) cells (a new immunotherapy)

INTERVENTIONS:
Other: Natural Killer (NK) cells (a new immunotherapy) — It is proposed to infuse allogeneic NK cells from a haploidentical donor, after administration of lymphoablative chemotherapy and/or radiotherapy, as a treatment in patients with sarcomas, who have completed conventional treatment but maintain detectable residual disease.
  The administration of low doses of radiotherapy is aimed at stressing residual tumor cells by increasing the expression of NK cell activating receptor ligands.
  The administration of prior chemotherapy aims at immunosuppressing the patient, allowing immunotherapy with allogeneic NK cells from haploidentical donor as well as autologous NK cell recovery to lead the immune reconstitution after chemotherapy, prolonging the antitumor effect.
  In conjunction with NK cell infusion, low doses (1x106/UI/m2) of interleukin 2 (IL-2) will be administered subcutaneously every 48h for a maximum of 6 doses, to favor the expansion and antitumor effect of NK cells.

SUMMARY:
This is an exploratory therapeutic study (according to the terminology of the "ICH Harmonised Tripartite Guideline Topic E8. General Considerations for Clinical Trials". EMEA, March 1998. CPMP/ICH/291/95), open-label, non-randomized, multicenter study. It is considered phase I/II since the safety and efficacy of the infusion of allogeneic haploidentical NK cells in combination with chemotherapy and/or radiotherapy in the treatment of pediatric, adolescent and young adult patients with refractory sarcoma will be sought.

DETAILED DESCRIPTION:
Metastatic or relapsed sarcoma in children, adolescents and young adults has a 5-year survival rate of less than 20% and current therapies, consisting of radical surgery and neoadjuvant chemotherapy, are ineffective and new therapeutic strategies are needed.

Natural Killer (NK) cell therapy is a new immunotherapy in development for cancer treatment. We propose a phase I/II clinical trial with the aim of determining the safety and efficacy of infusion of activated and expanded NK cells (NKAE) from a haploidentical donor in children suffering from sarcoma refractory to conventional therapy. The study will be carried out at Hospital Universitario La Paz (Madrid), Hospital Universitario Virgen de la Arrixaca (Murcia) and Hospital Universitario Cruces (Bilbao).

The results of this study are expected to have a direct influence on the approach to metastasis and refractoriness in pediatric solid tumors in future medical therapies.

It is expected to recruit 10 patients who, having received conventional treatment and/or salvage, continue to present metastatic disease or progression. Each patient will receive:

1. One cycle of lymphoablative chemotherapy: cyclophosphamide 60 mg/kg iv on day -6 and fludarabine 25 mg/m2/day iv on days -5 to -1.
2. Irradiation (2Gy) localized to the tumor and/or its metastases, ideally within 48h prior to NK cell infusion.
3. NK cells: Two infusions of cells separated by at least 4 days are established. The first infusion, day 0, will infuse up to 5x107/kg cells with NK and NKT immunophenotype (CD56+CD3- and CD3+). The first infusion will ideally be performed 24-48 h after completion of immunoablative chemotherapy. The second infusion, starting at day +4, up to 5x108/kg, provided that there has been no toxicity attributable to the infusion of the cell product in the previous cycle. In no case will more than 1x107/kg immunophenotype T cells (CD56-CD3+) be infused.
4. Cytokine IL-2: Starting on day -1 IL-2 will be administered at a dose of 1x106 IU/m2 subcutaneously every 48 hours, a total of 6 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 0 and 30 years diagnosed with malignant sarcoma, who at the end of conventional treatment still have detectable residual disease (based on imaging techniques) or in case of stable disease or minimal disease when there is an absence of clinical benefit from chemotherapy (poor tolerance due to adverse effects related to chemotherapy).
2. Lansky/Karnofsky index > 60%.
3. Mild-moderate (<4) organ functional impairment (hepatic, renal, respiratory), according to National Cancer Institute criteria (NCI CTCAE v5.0).
4. Left ventricular ejection fraction >39%.
5. Adult subjects who voluntarily signed informed consent prior to the first study intervention.
6. Minor subjects whose representative/legal guardian voluntarily signed the informed consent prior to the first intervention of the study.
7. In the case of mature minors (12 - 17 years of age), in addition to the consent signed by the legal guardian, the minor's assent will be obtained.
8. Women of childbearing capacity must have a negative pregnancy test at the time of inclusion and must agree to use highly effective contraceptive methods (diaphragms plus spermicide or male condom plus spermicide, oral contraceptive combined with a second method of contraceptive implant, injectable contraceptive, permanent intrauterine device, sexual abstinence or partner with vasectomy) during their participation in the study and within 30 days of the last visit.
9. Presence of a compatible haploidentical donor (father or mother or sibling).

Exclusion Criteria:

1. Patients with a history of poor therapeutic compliance.
2. Patients who, after a psycho-social evaluation, are censored as unsuitable for the procedure.

   * Socio-familial situation that makes proper participation in the study impossible.
   * Patients with emotional or psychological problems secondary to the disease, such as post-traumatic stress disorder, phobias, delirium, psychosis, requiring specialist support.
   * Evaluation of the involvement of family members in the patient's health.
   * Impossibility to understand information about the trial.
3. Severe functional organ impairment (hepatic, renal, respiratory) (4), according to the criteria of the National Cancer Institute (NCI CTCAE 5.0).
4. Contraindications, interactions, precautions for use and dose reductions indicated in the corresponding data sheets must be considered.
5. Subjects who have been administered other investigational drugs in the 90 days prior to inclusion.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2029-10-24 (Estimated); Study Completion 2029-10-24 (Estimated)

PRIMARY OUTCOMES:
Safety of allogeneic haploidentical adult differentiated Natural Killer cell infusion | Through study completion, an average of 7 years
  Safety of infusion of allogeneic haploidentical adult differentiated Natural Killers cells in combination with inteleukin-2 after chemotherapy and radiotherapy.
  Each patient will be monitored for the detection of possible adverse effects. The Common Terminology Criteria for Adverse Events V5.0 will be followed and the proportion of patients with toxicity will be determined according to the degree of toxicity. The intensity of toxic effects that cannot be classified according to the criteria for toxicity of the aforementioned system will be classified as follows (MedDRA classification):
  (a) Mild (asymptomatic); b) Moderate (symptomatic but does not significantly interfere with function); c) Severe (causes significant interference with function); d) Life-threatening

SECONDARY OUTCOMES:
Disease progression | Five-year after treatment
  Disease progression rate after treatment with Natural Killer (NK) + Inteleukin-2 (IL-2) cells will be determined by imaging techniques.
Infections (viral, fungal) | Through study completion, an average of 7 years
  Incidence of episodes of infections (viral, fungal) and hospital admissions associated with treatment.
Expression levels of Natural Killer cell inhibitory/activating ligands | Through study completion, an average of 7 years
  Expression levels of Natural Killer (NK) cell inhibitory/activating ligands in solid tumor samples and patient serum. These will be determined by immunohistochemistry and Polymerase Chain Reaction (PCR) techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No